CLINICAL TRIAL: NCT00166166
Title: Physiology and Pathologic Role of Endothelium-Derived Hyperpolarizing Factor in Humans
Brief Title: Endothelial Hyperpolarization in Humans
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited clinical staff
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00021886; 1R01HL079115-01 (NIH); 0605-2002 (Other: Other)
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Hyperlipidemia
Keywords: hyperlipidaemia; EDHF; FMD
MeSH Terms: conditions — Hyperlipidemias | interventions — Tetraethylammonium; omega-N-Methylarginine; Bradykinin; Nitroprusside; Acetylcholine; Sodium Chloride; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Controls (Experimental): Healthy subjects had venous occlusion plethysmography after intra-arterial infusions of saline, L-NG-monomethyl Arginine (L-NMMA), Tetraethylammonium (TEA), fluconazole, bradykinin, sodium nitroprusside and acetylcholine
  Interventions: Drug: Tetraethylammonium (TEA); Drug: L-NG-monomethyl Arginine (L-NMMA); Drug: Bradykinin; Drug: Sodium nitroprusside; Drug: Acetylcholine; Drug: Saline; Drug: Fluconazole
- Risk Factors (Experimental): Non-hypertensive subjects with cardiovascular risk factors had venous occlusion plethysmography after intra-arterial infusions of saline, L-NG-monomethyl Arginine (L-NMMA), Tetraethylammonium (TEA), fluconazole, bradykinin, sodium nitroprusside and acetylcholine
  Interventions: Drug: Tetraethylammonium (TEA); Drug: L-NG-monomethyl Arginine (L-NMMA); Drug: Bradykinin; Drug: Sodium nitroprusside; Drug: Acetylcholine; Drug: Saline; Drug: Fluconazole

INTERVENTIONS:
Drug: Tetraethylammonium (TEA) — 5 minute intra-arterial infusion of Tetraethylammonium at 1 mg/min
Drug: L-NG-monomethyl Arginine (L-NMMA) — 5 minute intra-arterial infusion of L-NMMA 8 μmol/min
  Other Names: Methylarginine
Drug: Bradykinin — Intra-arterial infusion of bradykinin at 100, 200, and 400 ng/min. Each dose will be given for 5 minutes.
Drug: Sodium nitroprusside — Intra-arterial infusion of sodium nitroprusside at 1.6 and 3.2 mg/min. Each dose will be given for 5 minutes.
  Other Names: Nitropress
Drug: Acetylcholine — Intra-arterial infusion of acetylcholine at 7.5, 15 and 30 μg/min. Each dose will be given for 5 minutes.
Drug: Saline — 5 minute intra-arterial infusion of 0.9% saline at 2.5ml/min
Drug: Fluconazole — 5 minute intra-arterial infusion of fluconazole at 0.4 mg/L/min
  Other Names: Diflucan

SUMMARY:
The purpose of this study is to elucidate the role Endothelium-Derived Hyperpolarizing Factor (EDHF) plays in dilating blood vessels and whether it differs between healthy people and those with high cholesterol. A second purpose of the study is to determine the identity of EDHF.

DETAILED DESCRIPTION:
The vascular endothelium synthesizes at least four potent vasodilator substances: nitric oxide (NO), prostacyclin, carbon monoxide and endothelium-derived hyperpolarizing factor (EDHF) that contribute to vasodilator tone, and to inhibition of platelet activation and inflammation. EDHF release is stimulated by receptor-dependent agonists such as acetylcholine and bradykinin (BK), and leads to hyperpolarization of the underlying smooth muscle cells presumably by opening Ca2+-activated K+ channels. Indirect pharmacological evidence suggests that EDHF is a cytochrome P450-derived arachidonic acid metabolite, presumably an epoxide. Although the pivotal role of NO to conduit vessel dilation in response to acute increases in shear stress is well known, its' contribution to dilation with sustained increases in flow are minimal, and may be due to EDHF release.

ELIGIBILITY:
Inclusion Criteria:

* Hyperlipidemic (LDL > 140)
* Healthy Volunteer

Exclusion Criteria:

* Pregnancy
* Diabetes mellitus
* Cardiovascular Disease
* Hypertension
* Use of any regular medications
* Renal insufficiency
* Smoking (current or within the past 5 years)
* Bleeding disorder

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2002-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arshed A Quyyumi, MD, Principal Investigator — Emory University School of Medicine, Division of Cardiology
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

REFERENCES:
- [Result] Ozkor MA, Murrow JR, Rahman AM, Kavtaradze N, Lin J, Manatunga A, Quyyumi AA. Endothelium-derived hyperpolarizing factor determines resting and stimulated forearm vasodilator tone in health and in disease. Circulation. 2011 May 24;123(20):2244-53. doi: 10.1161/CIRCULATIONAHA.110.990317. Epub 2011 May 9. PMID 21555712
- [Derived] Ozkor MA, Hayek SS, Rahman AM, Murrow JR, Kavtaradze N, Lin J, Manatunga A, Quyyumi AA. Contribution of endothelium-derived hyperpolarizing factor to exercise-induced vasodilation in health and hypercholesterolemia. Vasc Med. 2015 Feb;20(1):14-22. doi: 10.1177/1358863X14565374. Epub 2015 Feb 3. PMID 25648989
- [Derived] Rahman AM, Murrow JR, Ozkor MA, Kavtaradze N, Lin J, De Staercke C, Hooper WC, Manatunga A, Hayek S, Quyyumi AA. Endothelium-derived hyperpolarizing factor mediates bradykinin-stimulated tissue plasminogen activator release in humans. J Vasc Res. 2014;51(3):200-8. doi: 10.1159/000362666. Epub 2014 Jun 4. PMID 24925526
- [Derived] Ozkor MA, Rahman AM, Murrow JR, Kavtaradze N, Lin J, Manatunga A, Hayek S, Quyyumi AA. Differences in vascular nitric oxide and endothelium-derived hyperpolarizing factor bioavailability in blacks and whites. Arterioscler Thromb Vasc Biol. 2014 Jun;34(6):1320-7. doi: 10.1161/ATVBAHA.113.303136. Epub 2014 Mar 27. PMID 24675657

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Controls | Risk Factors
Started | 103 | 71
Completed | 103 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics represent subjects that completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Risk Factors | Total
Number analyzed (Participants) | 103 | 71 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11) | 46 (12) | 40 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 32 | 81
  Male | 54 | 39 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Forearm Blood Flow (FBF) After Tetraethylammonium (TEA) Administration
Description: Simultaneous forearm blood flow (FBF) measurements were obtained in both arms using a dual-channel venous occlusion strain gauge plethysmograph at rest and after administration of tetraethylammonium (TEA). Flow measurements were recorded for approximately 7 seconds, every 15 seconds up to eight times and a mean FBF value was computed. Percent change is the difference from baseline FBF and after TEA administration.
Time Frame: Baseline, 5 minutes
Population: Only 62 of the original 174 subjects were treated for this portion of the study.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Healthy Controls: Healthy subjects had venous occlusion plethysmography after intra-arterial infusions of saline (baseline) and Tetraethylammonium (TEA).
- Risk Factors: Non-hypertensive subjects with cardiovascular risk factors had venous occlusion plethysmography after intra-arterial infusions of saline (baseline) and Tetraethylammonium (TEA)
Arm/Group | Healthy Controls | Risk Factors
Number analyzed (Participants) | 37 | 25
percent change | -18 (16) | -24 (13)

2. Primary Outcome: Percent Change in Forearm Blood Flow (FBF) After Administration of L-NG-monomethyl Arginine (L-NMMA)
Description: Simultaneous forearm blood flow (FBF) measurements were obtained in both arms using a dual-channel venous occlusion strain gauge plethysmograph after administration of L-NG-monomethyl Arginine (L-NMMA). Flow measurements were recorded for approximately 7 seconds, every 15 seconds up to eight times and a mean FBF value was computed. Percent change is the difference in FBF from baseline and after L-NMMA administration.
Time Frame: Baseline, 5 minutes
Population: Only 62 of the original 174 subjects were treated for this portion of the study.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Healthy Controls: Healthy subjects had venous occlusion plethysmography after intra-arterial infusions of saline (baseline) and L-NG-monomethyl Arginine (L-NMMA)
- Risk Factors: Non-hypertensive subjects with cardiovascular risk factors had venous occlusion plethysmography after intra-arterial infusions of saline (baseline) and L-NG-monomethyl Arginine (L-NMMA)
Arm/Group | Healthy Controls | Risk Factors
Number analyzed (Participants) | 37 | 25
percent change | -29 (17) | -23 (15)

3. Secondary Outcome: Percent Change in Forearm Blood Flow (FBF) After Administration of L-NG-monomethyl Arginine (L-NMMA) and Tetraethylammonium (TEA)
Description: Simultaneous forearm blood flow (FBF) measurements were obtained in both arms using a dual-channel venous occlusion strain gauge plethysmograph after administration of L-NG-monomethyl Arginine (L-NMMA) and Tetraethylammonium (TEA). Flow measurements were recorded for approximately 7 seconds, every 15 seconds up to eight times and a mean FBF value was computed. Percent change is the difference in FBF from after L-NMMA administration and after TEA administration.
Time Frame: 5 minutes, 10 minutes
Population: Only 62 of the original 174 subjects were treated for this portion of the study.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Healthy Controls | Risk Factors
Number analyzed (Participants) | 37 | 25
percent change | -38 (17) | -39 (17)

4. Secondary Outcome: Percent Change in Forearm Blood Flow (FBF) After Fluconazole Administration
Description: Simultaneous forearm blood flow (FBF) measurements were obtained in both arms using a dual-channel venous occlusion strain gauge plethysmograph at rest and after administration of fluconazole. Flow measurements were recorded for approximately 7 seconds, every 15 seconds up to eight times and a mean FBF value was computed. Percent change is the difference from baseline FBF and after fluconazole administration.
Time Frame: Baseline, 5 minutes
Population: Only 33 of the original 174 subjects were treated for this portion of the study.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Healthy Controls: Healthy subjects had venous occlusion plethysmography after intra-arterial infusions of saline (baseline) and fluconazole.
- Risk Factors: Non-hypertensive subjects with cardiovascular risk factors had venous occlusion plethysmography after intra-arterial infusions of saline (baseline) and fluconazole
Arm/Group | Healthy Controls | Risk Factors
Number analyzed (Participants) | 26 | 7
percent change | -13 (16) | -17 (13)

5. Secondary Outcome: Percent Change in Forearm Blood Flow (FBF) After L-NG-monomethyl Arginine (L-NMMA) and Fluconazole Administration
Description: Simultaneous forearm blood flow (FBF) measurements were obtained in both arms using a dual-channel venous occlusion strain gauge plethysmograph after L-NMMA administration and administration of fluconazole. Flow measurements were recorded for approximately 7 seconds, every 15 seconds up to eight times and a mean FBF value was computed. Percent change is the difference in FBF after L-NMMA administration and then fluconazole administration.
Time Frame: 5 minutes, 10 minutes
Population: Only 15 of the original 174 subjects were treated for this portion of the study.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Healthy Controls: Healthy subjects had venous occlusion plethysmography after intra-arterial infusions of L-NG-monomethyl Arginine (L-NMMA), and fluconazole
- Risk Factors: Non-hypertensive subjects with cardiovascular risk factors had venous occlusion plethysmography after intra-arterial infusions of L-NG-monomethyl Arginine (L-NMMA) and fluconazole
Arm/Group | Healthy Controls | Risk Factors
Number analyzed (Participants) | 8 | 7
percent change | -26 (22) | -26 (22)

6. Secondary Outcome: Percent Change in Forearm Blood Flow (FBF) After Fluconazole and Tetraethylammonium (TEA) Administration
Description: Simultaneous forearm blood flow (FBF) measurements were obtained in both arms using a dual-channel venous occlusion strain gauge plethysmograph after administration of fluconazole and Tetraethylammonium (TEA) administration. Flow measurements were recorded for approximately 7 seconds, every 15 seconds up to eight times and a mean FBF value was computed. Percent change is the difference from FBF after fluconazole administration and after Tetraethylammonium (TEA) administration.
Time Frame: 5 minutes, 10 minutes
Population: Only 19 of the original 174 subjects were treated for this portion of the study.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Healthy Controls: Healthy subjects had venous occlusion plethysmography after intra-arterial infusions of fluconazole and Tetraethylammonium (TEA)
Arm/Group | Healthy Controls
Number analyzed (Participants) | 19
percent change | -22 (23)

7. Secondary Outcome: Forearm Blood Flow (FBF) After Sodium Nitroprusside Administration
Description: Simultaneous forearm blood flow (FBF) measurements were obtained in both arms using a dual-channel venous occlusion strain gauge plethysmograph after administration of sodium nitroprusside. Flow measurements were recorded for approximately 7 seconds, every 15 seconds up to eight times and a mean FBF value was computed.
Time Frame: 5 minutes
Population: Only 80 of the original 174 subjects were treated for this portion of the study.
Measure: Mean (Standard Error); unit: mL min^-1 * 100 mL^-1
Groups:
- Healthy Controls: Healthy subjects had venous occlusion plethysmography after intra-arterial infusions of sodium nitroprusside
- Risk Factors: Non-hypertensive subjects with cardiovascular risk factors had venous occlusion plethysmography after intra-arterial infusions of sodium nitroprusside
Arm/Group | Healthy Controls | Risk Factors
Number analyzed (Participants) | 42 | 38
mL min^-1 * 100 mL^-1 | 10.4 (4) | 10.9 (5)

8. Secondary Outcome: Change in Tissue Plasminogen Activator (t-PA) Release
Description: Individual net t-PA release at each time point were calculated by the following formula: net release = (Cv-CA) x {FBF x [101-hematocrit/100]}, where Cv and CA represent the concentration of t-PA in the brachial vein and artery, respectively. Change is the difference of t-PA at baseline and t-PA after bradykinin 400 ng/min
Time Frame: Baseline, 30 minutes
Population: Only 33 of the original 174 subjects were treated for this portion of the study.
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Healthy Controls: Healthy subjects had venous occlusion plethysmography after intra-arterial infusions of bradykinin
Arm/Group | Healthy Controls
Number analyzed (Participants) | 33
ng/mL | 5.6 (0.8)

9. Secondary Outcome: Change in Tissue Plasminogen Activator (t-PA) Release After Tetraethylammonium (TEA) and Bradykinin Administration
Description: Individual net t-PA release at each time point were calculated by the following formula: net release = (Cv-CA) x {FBF x [101-hematocrit/100]}, where Cv and CA represent the concentration of t-PA in the brachial vein and artery, respectively. Change is the difference of t-PA after Tetraethylammonium (TEA) and t-PA after bradykinin 400 ng/min
Time Frame: 30 minutes, 60 minutes
Population: Only 18 of the original 174 subjects were treated for this portion of the study.
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Healthy Controls: Healthy subjects had venous occlusion plethysmography after intra-arterial infusions of bradykinin and Tetraethylammonium (TEA)
Arm/Group | Healthy Controls
Number analyzed (Participants) | 18
ng/mL | 0.03 (0.7)

10. Secondary Outcome: Change in Tissue Plasminogen Activator (t-PA) Release After Fluconazole and Bradykinin Administration
Description: Individual net t-PA release at each time point were calculated by the following formula: net release = (Cv-CA) x {FBF x [101-hematocrit/100]}, where Cv and CA represent the concentration of t-PA in the brachial vein and artery, respectively. Change is the difference of t-PA after fluconazole and t-PA after bradykinin 400 ng/min
Time Frame: 30 minutes, 60 minutes
Population: Only 11 of the original 174 subjects were treated for this portion of the study.
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Healthy Controls: Healthy subjects had venous occlusion plethysmography after intra-arterial infusions of bradykinin and fluconazole
Arm/Group | Healthy Controls
Number analyzed (Participants) | 11
ng/mL | 4.4 (1.4)

11. Secondary Outcome: Change in Tissue Plasminogen Activator (t-PA) Release After Fluconazole, Tetraethylammonium (TEA), and Bradykinin Administration
Description: Individual net t-PA release at each time point were calculated by the following formula: net release = (Cv-CA) x {FBF x [101-hematocrit/100]}, where Cv and CA represent the concentration of t-PA in the brachial vein and artery, respectively. Change is the difference of t-PA after fluconazole and tetraethylammonium (TEA) and t-PA after bradykinin 400 ng/min
Time Frame: 60 minutes, 90 minutes
Population: Only 10 of the original 174 subjects were treated for this portion of the study.
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Healthy Controls: Healthy subjects had venous occlusion plethysmography after intra-arterial infusions of bradykinin, fluconazole and tetraethylammonium (TEA)
Arm/Group | Healthy Controls
Number analyzed (Participants) | 10
ng/mL | 1.6 (0.4)

ADVERSE EVENTS:
Arm/Group | Healthy Controls | Risk Factors
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/71
Other Adverse Events (participants affected / at risk) | 0/103 | 0/71

LIMITATIONS AND CAVEATS:
Findings are limited to the forearm microcirculations, thus other vascular beds including conductance arteries warrant further investigation. Nevertheless, it is known that the contribution of EDHF is less in conductance vessels than in microvessels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes